CLINICAL TRIAL: NCT03615430
Title: The Effect of Serratus Plane Block in Preventing Postoperative Pain and Chronic Pain After Breast Cancer Surgery
Brief Title: Serratus Plane Block in Preventing Postoperative Pain of Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Feng Xia (Other)
Responsible Party: Sponsor-Investigator, Feng Xia, Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2016]124
Record Dates: First submitted 2018-07-23; First posted 2018-08-03 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Serratus Plane Block; Chronic Pain; Breast Cancer
MeSH Terms: conditions — Chronic Pain; Breast Neoplasms | interventions — Anesthetics, Local; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): saline control group, 15 mL of the saline was administered to superficial and deep surface of serratus anterior in Control group via ultrasound before the surgery
  Interventions: Procedure: serratus plane block with saline
- SPB group (Experimental): Serratus plane block group, 15ml of 0.25% ropivacaine, a widely used local anesthetic for peripheral nerve block, was administered to superficial and deep surface of serratus anterior in SPB group via ultrasound before the surgery
  Interventions: Procedure: serratus plane block with local anesthetic

INTERVENTIONS:
Procedure: serratus plane block with local anesthetic — The high-frequency linear array ultrasound transducer (UST) was placed parallel to the cephalocaudal axis of the body in T4 levels on the side of the mid-axillary line, identifying latissimus dorsi and serratus anterior, through the thoracic artery to help to find the serratus anterior and 15 ml 0.25% ropivacaine was administered.
  Arms: SPB group
Procedure: serratus plane block with saline — The high-frequency linear array ultrasound transducer (UST) was placed parallel to the cephalocaudal axis of the body in T4 levels on the side of the mid-axillary line, identifying latissimus dorsi and serratus anterior, through the thoracic artery to help to find the serratus anterior and 15 ml saline was administered.
  Arms: Control group

SUMMARY:
A prospective, double-blinded randomized controlled, 1-year follow-up study was designed to compare the analgesic effect of serratus plane block (SPB) after breast cancer surgery. Women undergoing radical mastectomy were dIvided into Control group and SPB group. The postoperative acute pain was evaluated by numerical rating scale (NRS) and the effect of preventing chronic pain was assessed at 3, 6, 12 months after surgery by NRS.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing radical mastectomy with either sentinel lymph node dissection or axillary lymph node dissection or no axillary lymph node dissection
* between the ages of 18 and 85 yr
* with an American Society of Anesthesiology (ASA) physical status I or II
* without any significant cardiopulmonary, renal and hepatic dysfunction

Exclusion Criteria:

* Patients with any previous cancer other than breast cancer
* occurrence of allergy to local anesthetics
* occurrence of opioid-tolerant subjects
* occurrence of consuming analgesics, sedatives, antidepressants or any history of substance abuse before surgery

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — subject undergoing radical mastectomy
Enrollment: 50 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) of chronic pain | 3 months after surgery
  Pain intensity of patients was evaluated by Numerical Rating Scale, rating from 0 (no pain) to 10 (extreme pain) in order to evaluate the effect of SPB in preventing chronic pain

SECONDARY OUTCOMES:
the change trend of Numerical Rating Scale (NRS) after surgery | 0-24 hours after operation
  Pain intensity of patients was evaluated by Numerical Rating Scale, rating from 0 (no pain) to 10 (extreme pain) in order to evaluate the analgesic effect of SPB
Morphine consumption | 0-24 hours after operation
  extra need of analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Xia Feng, MD., Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Department of Anesthesiology, The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kamiya Y, Hasegawa M, Yoshida T, Takamatsu M, Koyama Y. Impact of pectoral nerve block on postoperative pain and quality of recovery in patients undergoing breast cancer surgery: A randomised controlled trial. Eur J Anaesthesiol. 2018 Mar;35(3):215-223. doi: 10.1097/EJA.0000000000000762. PMID 29227351